CLINICAL TRIAL: NCT03373721
Title: Gut Microbial Succession of Preterm Infants and Full-term Infants at Early Life
Brief Title: Gut Microbiota of Preterm Infants and Full-term Infants at Early Life
Status: Recruiting | Type: Observational
Sponsor: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: XH-17-009
Record Dates: First submitted 2017-12-11; First posted 2017-12-14 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Preterm Infant; Gut Microbiome
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Fecal samples of the recruited infants
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study is to obtain a longitudinal view of the gut microbial establishment of a cohort of 51 preterm (PT) infants compared to 50 full-term (FT) infants from birth to 90 days of age, and to identify key clinical factors that affect the establishment of neonatal microbiome.

The hypothesis of the investigators is that the gut microbiota progression of PT group and FT group is different in diversity and composition. Antibiotics and its usage duration is likely the main factor disturbing the colonization and development of the gut microbiome of PT infants.

DETAILED DESCRIPTION:
Premature birth is a global clinical problem. Early colonization and development of the neonatal gut microbiome is critically important with a profound impact on the host lifelong health. V3-V4 region of 16S rRNA amplicons of 581 stool DNA will be sequenced from a cohort of 51 PT infants and 50 FT infants to examine the microbial profiles. A random-effects generalized least square regression model is used to compare the difference in the main bacterial groups over time with the adjustment for multiple variables including gestational age and use of antibiotics .

ELIGIBILITY:
Inclusion Criteria:

Preterm infants

1. gestational age <37 weeks;
2. no gastrointestinal tract disorders, metabolic diseases, or viral hepatitis;
3. hospital stay > 7 days;

Exclusion criteria:

1. NICU stay less than 7 days
2. Necrotizing enterocolitis infant

Control group:

1. Full-term healthy infants;
2. gestational age >37 weeks;
3. vaginally born;
4. no gastrointestinal tract disorders, metabolic diseases, or viral hepatitis.

Ages: 1 Day to 4 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: About 50 preterm infants and 50 full-term healthy infants
Sampling Method: Probability Sample
Enrollment: 102 (Estimated)
Dates: Start 2014-07-20 (Actual); Primary Completion 2026-11-01 (Estimated); Study Completion 2028-12-20 (Estimated)

PRIMARY OUTCOMES:
changes in gut microbiota over time and in relation to antibiotic treatment | 0-7 years after birth
  Fecal DNA at different time points to measure the gut microbiota of preterm infants and full-term infants to investigate the development of early microbial colonization and the impact of antibiotics on the early life of preterm infants

CONTACTS AND LOCATIONS:
Overall Officials: Jie Jia, PhD, Principal Investigator — Xinhua Hospital, Shanghai Jiao Tong University School of Medicine
Locations (1):
- Department of NICU, XinHua Hospital Affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Jia J, Shuai M, Yan W, Tang Q, Wang B, Tang W, Wang P, Zhang T, Yang S, Zhang Y, Liu Q, Fu Y, Cai W, Zheng JS. Conserved Covarying Gut Microbial Network in Preterm Infants and Childhood Growth During the First 5 Years of Life: A Prospective Cohort Study. Am J Clin Nutr. 2023 Sep;118(3):561-571. doi: 10.1016/j.ajcnut.2023.07.019. Epub 2023 Jul 29. PMID 37517614